CLINICAL TRIAL: NCT02167555
Title: Characterization of Wild Blueberry Polyphenols Bioavailability and Kinetic Profile Over 24-hour Period
Acronym: WBB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-020
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Overweight; Obese; Healthy
Keywords: Wild Blueberries; Polyphenolics
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wild Bluberries (Active Comparator): Active Comparator
  Interventions: Dietary Supplement: Active Comparator
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Active Comparator — Wild Blueberry Beverage
  Other Names: Wild Blueberries
  Arms: Wild Bluberries
Dietary Supplement: Placebo Comparator — Placebo Beverage
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Primary objective is to characterize the relative bioavailability and kinetic profile of wild blueberry polyphenols over 24-hours period.

Secondary objective is to examine the relationship between bioavailability and kinetic profile of wild blueberry polyphenols on markers of chronic diseases.

DETAILED DESCRIPTION:
This study is a randomized, single blinded, 2-arm, within-subjects, placebo-controlled design utilizing a multiple sampling, repeated measures paradigm to characterize the bioavailability and kinetic profile of wild blueberry polyphenols.

A planned sample size of 12 will be enrolled into the study. This study will require one initial screening visit, one pre-study visit, and 2 study visits. This study will take approximately 3-4 weeks per subject to complete.

The initial screening visit will provide subject with the informed consent document and determine subject eligibility through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey relate to general eating, health, and exercise habits.

If willing and eligible to participate, a 3-day food record (2 weekdays and 1 weekend day) will be instructed at the Screening Visit and collected at the Pre-study visit to assess subjects' baseline dietary intake pattern. Subjects will be instructed to follow a strictly limited polyphenolic diet for 7 days prior to the study and throughout their participation time, while maintaining their usual diet pattern and physical activity, with counseling by staff investigator and/or Registered Dietitian. A dinner meal will be provided the day before the study visit to control the second meal effect from the food and beverage intake of the night before the study visit.

Subject will arrive at the center in a fasted state for at least 10 hours, well hydrated and rested. Each study visit will require blood draws throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a registered nurse will place a catheter in subject's arm for the purpose of multiple blood sample collections and take the initial blood draw in the fasting state. Subjects will be randomized to receive a placebo or wild blueberry beverage treatment based on randomized treatment sequences at 2 study visits along with 3 standard meals (breakfast, lunch and dinner). The sequences of receiving the beverage treatments at each visit will be randomly assigned to one of two of following sequences: placebo-wild blueberry or wild blueberry-placebo.

Each study visit will involve with blood samples collection at time points 0 (fasting), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hour (h) for assessment of change in plasma metabolites of wild blueberry polyphenols and influence of metabolic and inflammation markers. Also, urine samples will be collected prior to the study treatment as a baseline and all voids over 6 time periods, 0 to 2 h, 2 to 4 h, 4 to 6 h, 6 to 8 h, 8 to 10h and 10 to 24 h during each study visit to assess wild blueberry polyphenolic metabolites.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 years of age
* Body Mass Index (BMI) range from 25 to 33 kg/m2
* Nonsmoker
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, anti-inflammatory drugs, dietary supplements, etc…
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol
* Weight stable: not gained or lost weight +/- 5 kg in previous 3 months

Exclusion Criteria:

* Men and women who smoke
* Past smokers: abstinence for minimum 2 years
* Men and women with known or suspected food intolerance, allergies or hypersensitivity
* Men and women known to have/diagnosed with diabetes mellitus
* Men and women who have fasting blood glucose concentrations > 110mg/dL
* Men and women who have uncontrolled blood pressure >120 mmHg/80 mmHg
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc...
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating
* Taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplement, anti-inflammation, lipid lowering medication, blood pressure lowering medication, etc... Subjects may choose to go off dietary supplements (requires 30 days washout); e.g., fish oil, probiotics, etc...
* Men and women who have donated blood within 3 months of the Screening Visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
* Men and women who are vegans
* Substance (alcohol or drug) abuse within the last 2 years
* Excessive coffee and tea consumers (> 4 cups/d) and berry consumers (>2 cups fresh/day
* Men and women who do excessive exercise regularly or athlete
* Unstable weight: gained or lost weight +/- 5 kg in previous 3 months
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-01-08 (Actual); Study Completion 2016-01-19 (Actual)

PRIMARY OUTCOMES:
Changes in plasma and urine polyphenol metabolite concentrations over 24 hours after wild blueberry consumption with a high carbohydrate and high fat meal. | 24 hours
  To assess the kinetic profile and bioavailability of wild blueberry polyphenols when consume with a meal

SECONDARY OUTCOMES:
Changes in metabolic and inflammation markers over 24 hours after wild blueberry consumption with a high carbohydrate and high fat meal. | 24 hours
  The influence of wild blueberry consumption on metabolic and inflammation markers

OTHER OUTCOMES:
Changes in oxidative stress markers over 24 hours after wild blueberry consumption with a high carbohydrate and high fat meal | 24 hours
  The influence of wild blueberry consumption on oxidative stress markers

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, MS, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhong S, Sandhu A, Edirisinghe I, Burton-Freeman B. Characterization of Wild Blueberry Polyphenols Bioavailability and Kinetic Profile in Plasma over 24-h Period in Human Subjects. Mol Nutr Food Res. 2017 Dec;61(12). doi: 10.1002/mnfr.201700405. Epub 2017 Nov 8. PMID 28887907